CLINICAL TRIAL: NCT01043939
Title: A Pilot Study to Evaluate the Effects of Purple Grape Juice on the Vascular Health of Childhood Cancer Survivors
Brief Title: Purple Grape Juice in Improving Vascular Health in Childhood Cancer Survivors
Acronym: JAVA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009NTLS074; NCI-2009-01497 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Disease
Keywords: childhood cancers; cardiovascular disease; childhood cancer survivor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purple Grape Juice First (Active Comparator): After 4 week run-in period, drink 6 ounces of purple grape juice twice daily, then 4 week washout, week 12 drink 6 ounces of clear apple juice for 4 weeks twice daily
  Interventions: Other: Purple Grape Juice; Other: Apple Juice
- Apple Juice First (Active Comparator): After 4 week run-in period, drink 6 ounces of clear apple juice twice daily, then 4 week washout, week 12 drink 6 ounces of purple grape juice for 4 weeks twice daily
  Interventions: Other: Purple Grape Juice; Other: Apple Juice

INTERVENTIONS:
Other: Purple Grape Juice — 6 ounces of purple grape juice consumed twice daily either during first or second 4 week supplementation period, depending on sequence randomization
Other: Apple Juice — 6 ounces of clear apple juice consumed twice daily either during first or second 4 week supplementation period, depending on sequence randomization
  Other Names: clear apple juice

SUMMARY:
Rationale: Survivors of childhood cancer are at an increased risk of developing cardiovascular risk factors as well as early cardiovascular disease, likely due to the intensive therapeutic regimen used to treat their cancer. Purple grape juice (PGJ) is a rich source of flavonoids and a powerful antioxidant. Clinical studies in both diseased and healthy adults suggest that daily consumption of PGJ contributes to increased antioxidant capacity, reduced low-density lipoprotein (LDL) oxidation, and improved vasodilation.

Purpose: This randomized clinical trial is evaluating whether purple grape juice can reduce oxidative stress and improve the vascular health of survivors of childhood cancer in the early stages of cardiovascular disease.

DETAILED DESCRIPTION:
Primary Objective:

* To evaluate the effect of PGJ on endothelial function, a key measure of vascular health and considered a barometer for cardiovascular disease risk.

Secondary Objective:

* To evaluate the effect of PGJ on biomarkers of vascular and systemic oxidative stress.

Outline:

Patients undergo a 4-week washout period and refrain from consuming any type of juice, juice drink (less than 100% juice), wine or grapes. Patients are then randomized to 1 of 2 arms.

Arm 1: Beginning in week 4, patients consume 6 ounces of purple grape juice (PGJ) twice daily for 4 weeks. Beginning in week 12, after a 4 week washout period, patients crossover to consume apple juice (AJ) as in Arm 2.

Arm 2: Beginning in week 4, patients consume 6 ounces of AJ twice daily for 4 weeks. Beginning in week 12, after a 4 week washout period, patients crossover to consume PGJ as in Arm 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer > 5 years ago
* Off-maintenance therapy for > 36 months
* Age 10-30 years
* Reside within a 50 mile radius of the University of Minnesota

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Start of oral contraceptives < or = 3 months prior to study enrollment
* Current smoker
* Diabetes (type 1 and 2)
* Antibiotic use < 2 weeks prior to study enrollment

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Blair, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Minnesota General Clinical Research Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Metabolic Syndrome Study in Childhood Cancer Survivors and the Long-Term Follow-up Clinic, both at the University of Minnesota, Minneapolis, MN between October 2009 and May 2010.
Pre-assignment Details: 30 recruited; 6 drop-outs during 4 week run-in period, prior to randomization due to now-show for first clinic visit or concerns regarding time, compliance, or blood draws.
Groups:
- Arm 1 Purple Grape Juice Then Apple Juice: Arm 1: 6 ounces of grape juice twice daily during first 4 weeks of intervention (intervention period 1) followed by a 4 week washout period followed by 6 ounces of clear apple juice twice daily during 4 weeks (intervention period 2).
- Arm 2 Apple Juice Then Purple Grape Juice: Arm 2: 6 ounces of clear apple juice twice daily during first 4 weeks of intervention (intervention period 1) followed by a 4 week washout period followed by 6 ounces of purple grape juice twice daily during 4 weeks (intervention period 2).
Period: First Intervention
Arm/Group | Arm 1 Purple Grape Juice Then Apple Juice | Arm 2 Apple Juice Then Purple Grape Juice
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Arm 1 Purple Grape Juice Then Apple Juice | Arm 2 Apple Juice Then Purple Grape Juice
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Arm 1 Purple Grape Juice Then Apple Juice | Arm 2 Apple Juice Then Purple Grape Juice
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive purple grape juice first and apple juice first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 24
Weight [Mean (Standard Deviation); unit: kilograms] — Measured in kilograms at beginning of study.
  kilograms | 60 (13.8)
Height [Mean (Standard Deviation); unit: Centimeters] — Measured in centimeters are beginning of study.
  Centimeters | 165 (11.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Measured in kilograms/m^2 at beginning of study.
  kg/m^2 | 22 (3.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 111 (9.6)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 59 (8.3)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 78 (7.0)
Fasting insulin [Mean (Standard Deviation); unit: mU/L] | 6.3 (4.7)
Low-density lipoprotein (LDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 95 (20.1)
High-density lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 50 (10.9)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 78 (33.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Function (Reactive Hyperemia Peripheral Arterial Tonometry (RH-PAT) Index Score)
Description: Difference of least square means (95% Confidence Interval) in RH-PAT Index Scores between juice groups. Higher RH-PAT scores indicate better endothelial function; a positive difference of least square means is suggestive of an improvement in endothelial function.
  Probes were placed on the index fingers of both hands and a blood pressure cuff was placed on one arm. The cuff was inflated to suprasystolic pressure and the digital pulse volume was recorded before, during & after a 5 minute occlusion period. The ratio of the hyperemic and the baseline pulse amplitude (corrected for the same ratio on the control finger) was calculated and expressed as the RH-PAT index score. Lower scores reflect worse endothelial function.
Time Frame: 4 weeks (change since baseline)
Population: Intent-to-Treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Purple Grape Juice: 6 ounces of grape juice consumed twice daily in either the first or second intervention period
- Apple Juice: 6 ounces of clear apple juice consumed twice daily in either the first or second intervention period
Arm/Group | Purple Grape Juice | Apple Juice
Number analyzed (Participants) | 24 | 24
units on a scale | 0.06 (0.089) [-0.42 to 0.11] | 0.22 (0.093) [-0.42 to 0.22]
Statistical Analysis 1: Comparison: Purple Grape Juice vs Apple Juice; Test type: Superiority or Other; p = 0.25, Mixed Models Analysis — 24 participants required to achieve 80% power to detect mean difference of 0.3 in RH-PAT index score between juice groups, assuming standard deviation of the difference was 0.25, using a two-sided significance level of 0.05; Mixed effects ANCOVA model with baseline included as a covariate, subject as a random effect; juice, period & group as fixed effects; Difference of least square means = -0.16, 95% CI 2-sided [-0.42 to 0.11] — The a priori threshold for statistical significance was 0.05

2. Secondary Outcome: Change in Oxidized LDL
Description: Change from baseline in Oxidized LDL at 4 weeks, a biomarker of oxidative stress
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Units/Liter
Arm/Group | Purple Grape Juice | Apple Juice
Number analyzed (Participants) | 24 | 24
Units/Liter | 4.66 (2.02) | 1.57 (2.03)
Statistical Analysis 1: Comparison: Purple Grape Juice vs Apple Juice; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Difference of least square means = 3.09, 95% CI 2-sided [-2.73 to 8.91]

3. Secondary Outcome: Change in Myeloperoxidase (MPO)
Description: Change from baseline in Myeloperoxidase (MPO) at 4 weeks, a biomarker of oxidative stress
Time Frame: 4 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Arm 2 Apple Juice Then Purple Grape Juice: 6 ounces of clear apple juice consumed twice daily in either the first or second intervention period
Arm/Group | Purple Grape Juice | Arm 2 Apple Juice Then Purple Grape Juice
Number analyzed (Participants) | 24 | 24
ng/mL | 0.95 [0.78 to 1.16] | 1.03 [0.84 to 1.26]
Statistical Analysis 1: Comparison: Purple Grape Juice vs Arm 2 Apple Juice Then Purple Grape Juice; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of means = 0.92, 95% CI 2-sided [0.82 to 1.03] — MPO was log transformed prior to analyses; the difference of log-transformed least square means (95% CI) were back-transformed to obtain the ratio of the means (95% CI)

4. Secondary Outcome: Change in High Sensitivity C-Reactive Protein (Hs-CRP)
Description: Change from baseline in high sensitivity C-Reactive Protein (hs-CRP) at 4 weeks, a biomarker of inflammation
Time Frame: 4 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Purple Grape Juice | Apple Juice
Number analyzed (Participants) | 24 | 24
mg/L | 1.42 [0.84 to 2.41] | 1.06 [0.62 to 1.80]
Statistical Analysis 1: Comparison: Purple Grape Juice vs Apple Juice; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio of means = 1.34, 95% CI 2-sided [0.69 to 2.62] — hs-CRP was log transformed prior to analyses; the difference of log-transformed least square means (95% CI) were back-transformed to obtain the ratio of the means (95% CI)

ADVERSE EVENTS:
Arm/Group | Purple Grape Juice | Apple Juice
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes